CLINICAL TRIAL: NCT01735357
Title: Investigation Into Incorporation of (n-3) Polyunsaturated Fatty Acids Into Erythrocyte Membranes and Clearance, and Effects on Platelet Function, Arterial Function and Endothelial Repair
Brief Title: Differential Effects of Eicosapentaenoic Acid (EPA) and Docosahexaenoic Acid (DHA) on Platelet, Endothelial and Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Dr Wendy Hall, Lecturer in Nutritional Sciences, King's College London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EDT
Record Dates: First submitted 2012-11-20; First posted 2012-11-28 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Healthy
Keywords: Eicosapentaenoic acid; Docosahexaenoic acid; Cardiovascular risk; Platelet function; Endothelial function; Vascular function; young males

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Olive oil (BP specification) (Placebo Comparator): 5g per day
  Interventions: Dietary Supplement: Placebo - olive oil (BP specification)
- DHA-rich oil (Experimental): Fish oil supplement (total = 5g/day) providing 3.1g/day of DHA triacylglycerol, blended with olive oil
  Interventions: Dietary Supplement: DHA-rich triacylglycerol oil
- EPA-rich oil (Experimental): Fish oil supplement (total = 5g/day) providing 2.9g/day of EPA triacylglycerol, blended with olive oil
  Interventions: Dietary Supplement: EPA-rich triacylglycerol oil

INTERVENTIONS:
Dietary Supplement: EPA-rich triacylglycerol oil
  Arms: EPA-rich oil
Dietary Supplement: Placebo - olive oil (BP specification)
  Arms: Olive oil (BP specification)
Dietary Supplement: DHA-rich triacylglycerol oil
  Arms: DHA-rich oil

SUMMARY:
The purpose of this study was to determine whether supplementation with oils enriched with long chain n-3 PUFA, either EPA or DHA, had a differential effect on platelet, endothelial and vascular function.

DETAILED DESCRIPTION:
Relatively few studies have made a head-to-head comparison of DHA (22:6n-3) with EPA (20:5n-3). The understanding of this differential effect may be of great interest in populations with low EPA intake such as vegetarians, who may choose to supplement their dietary intake of long-chain n-3 PUFA in the form of DHA-rich algal oil.

This study aimed to investigate the effect of supplementation with oils rich in either EPA or DHA (3g/day, 6 weeks) in healthy young males on platelet, endothelial and vascular function, as well as other CVD risk factors. The primary outcomes were platelet monocyte aggregates and endothelial progenitor cells - novel markers of platelet and endothelial function, measured by flow cytometry, Secondary outcomes included capillary density, measured by capillaroscopy to assess changes in microvascular function, pulse wave analysis, digital volume pulse and ambulatory blood pressure. Other secondary outcomes included lipid profiles (TAG, cholesterol, NEFA), glycaemic control (HOMA, QUICKI) and oxidative stress (isoprostane). The omega-3 index (erythrocyte EPA+DHA) was used as a marker of compliance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* No smokers
* Aged 18-45y old
* Able to understand the information sheet and comply with all the trial procedures
* Having given written consent to take part in the study prior to participation.

Exclusion Criteria:

* Reported history of CVD (myocardial infarction, angina, venous thrombosis, stroke, dyslipidemia), diabetes (or fasting glucose ≥ 6.1 mmol/L), cancer, kidney, liver or bowel disease.
* Presence of gastrointestinal disorder or use of drug, which is likely to alter gastrointestinal motility or nutrient absorption.
* Current smokers; history of substance abuse or alcoholism (previous weekly alcohol intake >60 units/week); current self-reported weekly alcohol intake exceeding 28 units
* Recent use of hypolipidaemic, antihypertensive, antiplatelet or antithrombotic mediations
* Platelet count above or below the normal range or any history indicative of a congenital or acquired platelet or haemostatic defect.
* Allergy or intolerance to any component of study capsules
* Unwilling to restrict consumption of any source of fish oil for the length of the study
* Subjects reporting consumption of >1 portion oily fish per week
* Weight change of >3 kg in preceding 2 months; BMI <18 and >32 kg/m2
* Blood pressure>160/90 mmHg
* Fasting blood cholesterol > 6.5 mmol/L; fasting triacylglycerol concentrations > 2.0 mmol/L

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Platelet Monocyte Aggregates (PMA) | 6 weeks
  The endothelium plays a vital role in the regulation of blood flow, thrombosis and inflammation. Endothelium-derived anti-adhesive and anti-aggregant substances, including prostacyclin and nitric oxide, are known to inhibit platelet activation. Endothelial dysfunction or vessel wall injury lead to the activation of platelets, of which platelet-monocyte-aggregates (PMA) are a sensitive marker, and were shown to inversely correlate with markers of EF in patients with stable CHD. The measurement of PMA by flow cytometry is a method which reduces ex vivo platelet activation to its minimum and is believed to represent platelet activation in vivo.
Endothelial Progenitor Cell (EPC) counts | 6 weeks
  EPCs are a subgroup of circulating progenitor cells that are recruited from the bone marrow to repair the injured vasculature. They have been associated with a reduced CVD risk and may serve as markers of endothelial function because they represent a greater capacity for the endothelium to repair itself. Two populations of EPCs were measured by flow cytometry, described as 'early EPC' (KDR+/CD34+/CD133+) and 'late EPCs' (KDR+/CD34+/CD31+).

SECONDARY OUTCOMES:
Capillary density | 6 weeks
  Capillary rarefaction has been associated to CVD risk factors such as hypertension, smoking and obesity. The cutaneous circulation has emerged as an accessible and representative vascular bed to look at microvascular dysfunction. Capillary density was measured by a Capiscope (kk technologies)
Arterial stiffness | 6 weeks
  Pulse wave analysis (PWA) was used to measure indices of arterial stiffness, including peripheral and central augmentation index, as well as central systolic and diastolic blood pressure. Digital volume pulse (DVP) was used to measure reflection and stiffness indices.
Blood Pressure (BP) and Heart Rate (HR) | 6 weeks
  Resting HR and BP were measured in the seated and supine position after 15 minute rest, on the days of both baseline and endpoint visits. In addition, ambulatory BP and HR (24h, daytime, nighttime) was measured 2-3 days prior to each visit.
Plasma isoprostane concentrations | 6 weeks
  8-iso-prostaglandin-F2α (8-IsoP-F2α), a prostaglandin F2-like compound biosynthesized nonenzymatically by a free-radical oxygenation of arachidonic acid, was measured in plasma in order to assess oxidative stress.
Plasma Nitrate and Nitrites (NOx) concentrations | 6 weeks
  Plasma NOx was measured as a circulating marker of endothelial function.
Serum total cholesterol concentration | 6 weeks
Serum Triacylglycerol concentrations | 6 weeks
Serum high density lipoprotein concentration | 6 weeks
Serum low density lipoprotein concentration | 6 weeks
Serum non esterified fatty acids (NEFA) concentration | 6 weeks
Serum Apolipoprotein B concentration | 6 weeks
Plasma glucose concentration | 6 weeks
Plasma insulin concentration | 6 weeks
Serum adiponectin concentration | 6 weeks
Serum resistin concentration | 6 weeks
Erythrocyte phospholipid fatty acid profiles | 6 weeks
  The EPA and DHA content of erythrocyte lipids were used as a marker of compliance.
Fatty acid profile of plasma non esterified fatty acid fraction | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wendy L Hall, PhD, Principal Investigator — King's College London
Locations (1):
- Diabetes & Nutritional Sciences Division, King's College London, London, United Kingdom

REFERENCES:
- [Derived] Cottin SC, Alsaleh A, Sanders TA, Hall WL. Lack of effect of supplementation with EPA or DHA on platelet-monocyte aggregates and vascular function in healthy men. Nutr Metab Cardiovasc Dis. 2016 Aug;26(8):743-51. doi: 10.1016/j.numecd.2016.03.004. Epub 2016 Mar 15. PMID 27105870
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/27105870